# Developing Process-Specific Verbal Memory Interventions for Veterans with TBI

Protocol

NCT02310633

March 4, 2019

#### **Protocol**

- 1. Project Title: Developing Process-Specific Verbal Memory Interventions in Veterans with TBI
- 2. Investigator(s): Russell M. Bauer, Ph.D., Thomas Mareci, Ph.D., Mingzhou Ding, Ph.D.
- 3. Abstract: Memory dysfunction can result from impairments along a continuum of information processing, from poor initial acquisition of information during learning to disturbed retrieval of stored memory when it is later needed to perform a task<sup>1</sup>. There is a critical need to better understand disease heterogeneity in order to enhance diagnosis and therapeutic management<sup>2</sup>. Several subtypes of memory dysfunction after TBI have been identified<sup>3,4</sup>. First, some TBI survivors exhibit impaired memory acquisition/encoding (e.g., frontal system damage)<sup>5</sup>. Second, some exhibit impaired memory consolidation/storage impairment (e.g., prominent damage to temporal lobe systems<sup>6</sup>). Third, some show impairment in retrieval of information<sup>5,7</sup>. This heterogeneity results from the variable nature and severity of underlying brain trauma resulting from unpredictable mechanical forces<sup>2,8</sup>. This study attempts to determine whether these subtypes of memory respond better to treatments that are focused specifically on the constituent cognitive deficit than to other treatments. There are existing training protocols for training these three components of memory processing, as follows: encoding (memory strategy training<sup>9</sup>), consolidation (errorless learning<sup>10</sup>), and retrieval (retrieval practice<sup>11</sup>, but their efficacy has not been tested in TBI survivors with documented impairments in each component. That is, to our knowledge, there is no solid evidence for memory training in TBI survivors that supports the widely held belief that specifically matching the patient impairment to the treatment leads to better treatment outcomes. This project attempts to fill this gap in our knowledge. In an alternating treatments design, TBI survivors with encoding, consolidation, or retrieval deficits will undergo (a) a treatment matched to their deficit and (b) a treatment that addresses a different deficit. High resolution imaging and neurocognitive biomarkers will be used to predict response to treatment. Results will be used as a basis for a larger clinical trial of memory rehabilitation in brain injured populations.

### 4. Background:

Traumatic brain injury (TBI) has emerged as a "signature injury" of the OIF-OEF-OND combat experience. Enduring cognitive deficits after TBI present barriers to full recovery and re-entry into societal roles, with executive dysfunction, poor attention-concentration, and memory difficulties being the most persistent disabilities faced by TBI survivors<sup>12</sup>. Current Knowledge. There is considerable heterogeneity in the nature and severity of memory disorders after moderate-severe TBI(M-STBI)<sup>8</sup>, resulting not only from variability in severity and etiology of TBI, but also from variable loci of neuroanatomic damage<sup>13</sup>. Chronic episodic memory deficits after M-STBI are often rooted in deficient encoding and/or consolidation of tobe-learned information<sup>5,14</sup>, or from retrieval deficits associated with frontal-executive damage<sup>4</sup>. Meta-analytic reviews of memory rehabilitation studies show that memory strategy training may improve TBI-related memory deficits of any severity, leading to its recommendation by ACRM as a practice standard<sup>15</sup>. More limited data on errorless learning (EL), which rebuilds learning/memory skills in a way that prevents errors, suggests that EL is a promising approach to treating severe memory deficits<sup>10,16,17</sup>. Retrieval practice (in which participants practice the act of retrieving information with appropriate cueing and support) improves paired-associate

learning in the TBI population<sup>18,19</sup>. Other memory therapies with promising but unproven efficacy in RCT's include spaced retrieval<sup>20,21</sup> and the method of vanishing cues<sup>22,23</sup>. Gaps in Knowledge. Although these protocols may lead to improved learning and memory after M-STBI, little is known about their mechanism(s) of action or whether they would be differentially effective in TBI survivors with deficits at different stages of the memory process. There have been no comparative effectiveness studies involving these treatments, and no group studies have attempted to match patients to treatments that specifically target the locus of memory impairment in encoding, consolidation, or retrieval. If, in fact, some patients suffer from consolidation failure<sup>6</sup>, while others have prominent encoding or retrieval deficits<sup>5,24,25</sup>, it is likely that alternative memory interventions, each matched to the patient's primary deficit, may be needed to maximize individual rehabilitation outcomes. Stage of recovery/time since injury may also be important, as encoding deficits and consolidation deficits recover differentially in severely injured patients, with poor encoding representing the more enduring problem<sup>13</sup>. Relevance: Managing and alleviating residual effects of traumatic brain injury is a key priority area and represents a critically important public health problem facing the veteran population. Differential efficacy of specific rehabilitation programs may be an important factor for clinicians to consider when offering health services to veterans with cognitive impairment. Benefit to Veterans. A better understanding of the efficacy of memory rehabilitation may provide clinicians with better decision-making support for prescribing different available therapies to alleviate TBI-related cognitive and memory dysfunction. Better understanding of individual differences in TBI-related memory dysfunction, and of underlying structural and

### 5. Specific Aims:

difficulties veterans suffer after M-STBI.

<u>Aim 1.</u> Aim 1 is to refine and validate three separate, process-specific memory rehabilitation treatments that focus on improving information-processing at the encoding, consolidation, or retrieval stage for Veterans with chronic moderate/severe TBI.

functional brain dysfunction may also explain the neural basis for heterogeneous memory

Objective 1.1. Generate treatment manuals for three process-specific memory treatments. Objective 1.2. Test and refine treatment fidelity so that each of the three interventions can be reliably delivered by different clinicians.

<u>Aim 2.</u> Aim 2 is to provide a preliminary test of the response to the three memory interventions. At baseline, TBI survivors will be evaluated for memory function in each of these three memory component processes using established neuropsychometric methods. Their experimental treatment allocation will be to the treatment targeting their most impaired memory component. In addition, each subject will serve as his/her own control, by engaging in a treatment targeted to another memory component ('mismatched' group).

<u>Hypothesis A.</u> The <u>matched vs.</u> mismatched group will show differential improvement in memory component function, with the former group benefitting to a significantly greater degree. (Primary measures: Memory component performance, encoding, consolidation, retrieval; secondary: cognitive function and quality of life).

<u>Aim 3.</u> Aim 3 is to establish links between the behavioral taxonomy of the three memory components and differences in brain structure and function documented with diffusion tensor imaging and functional connectivity analysis. This is a key first step in establishing brain-based metrics of neuroplastic change after memory therapy in our research program.

Objective 3.1. Identify specific and unique imaging signatures that distinguish patients with deficits in encoding, consolidation, and retrieval, respectively. Primary measures: structural measures of morphometry and white matter integrity (FA) and functional connectivity (cross correlation and total interdependence) in identified brain networks damaged in TBI.

**Clinical Implications**. This research has the potential to devise a method to match specific

subcomponents of memory impairment to specifically targeted memory interventions, thus maximizing recovery of memory and function. The results of this investigation will be used to refine the interventions, to evaluate cognitive and functional endpoints, and to power a larger clinical trial that will yield data enabling clinicians to match TBI patients to effective treatments based on their individual profile of memory dysfunction.

# 6. Research Plan:

- **6.1.** <u>Study Design</u>. The proposed research will be conducted in three phases: Intervention Development, Patient Characterization and Classification, and Initial Testing of Treatment Efficacy.
- **6.2.** Phase 1: Intervention Development. During the first 6 months of the project, we will formalize, manualize, and perform preliminary fidelity testing on three memory interventions targeting process-specific memory deficits after TBI in Veterans: (a) memory strategy training (to boost encoding), (b) errorless learning (to improve consolidation, and (c) retrieval practice (to rehabilitate deficits in retrieval).
- 6.2.1. Materials Common to Memory Interventions. Each of the three treatment conditions will utilize the same training materials, a set of verbal paired-associates (VPA) and a set of face-name pairs (FNP), both presented for training in associative learning. Each session will involve training utilizing two 12-item VPA lists and two sets of 12 FNP's, for an overall total of 144 unique VPAs and 144 FNPs. The VPA's are weak paired associates<sup>26,27</sup> (have a forward association strength of <.01<sup>28</sup>), and that do not contain words from clinical memory tests given in Phase 2. FNP's are constructed by pairing face-front black and white photographs from Stringer's Ecologically-Oriented Neurorehabilitation of Memory (EON-MEM) protocol<sup>29</sup>. Training stimuli will be presented on a desktop computer using E-prime software.
- 6.2.2. Memory Strategy Training (MST). MST, in which persons with brain injury are taught specific strategies useful for encoding new information at the point of learning, is a widely used rehabilitative technique<sup>9,30,31</sup> that is an *ACRM practice standard*<sup>15</sup>. While specific strategies vary across studies, most teach the participant to form meaningful cognitive associations between memoranda through the use of imagery or semantic encoding, building a form of memory encoding known as relational memory<sup>32</sup>. Relational encoding, a key process that enhances the strength and durability of episodic memory<sup>33,34</sup>, can be reduced or impaired after TBI<sup>35</sup>. Successful relational memory involves two distinct mnemonic mechanisms: the generation of an association between to-be-encoded items (a frontal/executive function)<sup>36,37</sup> and the binding of that association into a cohesive memory trace (a function of the hippocampal memory system)<sup>33,38</sup>. MST may be particularly useful in enhancing the first of these two processes.
- 6.2.2.1. <u>Procedure</u>. Six biweekly sessions of MST will be conducted. Two VPA lists and two FNP lists will be used in each session. During MST, VPAs (e.g., "candle-table") or FNPs will be presented in horizontal arrangement on a computer screen at a rate of 1 per 6 seconds (this may be modified based on participant processing speed). For **VPA learning**, participants will be asked to generate a memorable sentence (first list) or form a distinctive mental image (second list) that links the two VPA items together. The therapist will help the participant generate sentences and images that are distinctive or unusual, and therefore more memorable. Specific examples of distinctive sentence-based and imagery-based encoding will be given (e.g., "The wax from the candle poured onto the table", or an image of a candle scorching a table) and will be developed as the treatment is manualized. Immediately following list presentation, the cue word will be presented without the target (e.g., "candle-\_\_\_\_\_\_") and the participant will be asked to generate the target. Spontaneous production of targets will be recorded. For each item not spontaneously recalled, participants will be asked to retrieve the

sentence (first list) or image (second list) that they created during encoding, and will then be asked to retrieve the target word again. Unsuccessful retrieval will be initially cued by the therapist. Prompted recall will also be recorded. This procedure will be repeated five times for each list, each followed by a retrieval phase. For each session, the dependent measure is the percentage of correct target words (out of 12) in spontaneous and cued recall for each list during the final exposure trial. For *FNP learning*, we will use a training approach adapted from Hampstead<sup>39</sup> and Stringer<sup>9</sup>. Training teaches patients to self-generate cues linking faces and names; patients will also be provided cues to standardize procedures and to encourage strategy development. For each FNP, participants will be directed to a salient facial feature (a visual cue like a long nose) and given a nickname that rhymes with the actual name (verbal cue) linking the feature to the name. Patients will be instructed to associate the visual and verbal cues by creating mental images that emphasize or exaggerate the relationship between cues. After initial learning, FNP's will be repeated five times. On each presentation, participants will be asked to recall the visual cue, then the verbal cue, and then finally the name. Dependent measure is the percent correct recall of visual cues, verbal cues, and names on the final trial of each list.

- 6.2.3. <u>Errorless Learning (EL).</u> EL refers to a group of techniques that promote recovery of memory abilities using procedures that explicitly prevent the patient from making errors during learning<sup>10</sup>. EL is based on the premise that errors during training become primed in long term memory via implicit memory mechanisms relatively spared in amnesia<sup>40</sup>. Because of impairment in explicit memory consolidation that would normally provide corrective influence, these errors exert an unusually strong detrimental effect on relearning. While the standard interpretation of EL is that implicit memory is responsible for the treatment effect<sup>41,42</sup>, it has been more recently shown that the EL advantage results from residual, though impaired, episodic memory consolidation due to temporal lobe damage<sup>43,44</sup>. EL has been shown to be a promising tool in memory rehabilitation<sup>15,40,45</sup>, at least for individuals without severe executive deficits<sup>46</sup>.
- 6.2.3.1. <u>Procedure</u>. Six biweekly sessions of EL will be conducted, each using two VPA lists and two FNP lists. During EL, the word pairs (e.g., "candle-table") or face-name pairs will be presented in horizontal arrangement on a computer screen at a rate of 1 per 6 seconds with no encoding instructions. After initial presentation, the cue will be presented without the target. For VPA learning, the cue word in each pair ("candle \_\_\_\_\_\_") will be presented, and the participant will be asked to provide the second (target) word, *but only if they are certain they can retrieve it accurately. Guessing is explicitly discouraged*. If the participant cannot provide the word within 3 seconds, the word appears on the screen for 3 seconds and the participant is asked to read the pair aloud. During training, each list will be presented five times in this fashion. The <u>dependent measure</u> is the percent correct target words produced (out of 12) during the fifth exposure trial for each list. The procedure will be repeated for the second VPA list and then for the two FNP lists, yielding 4 accuracy measures (percent correct) for each session.
- 6.2.4. Retrieval Practice (RP). Some authors have argued that practicing retrieval during learning is an essential feature of successful learning<sup>10,47</sup>. Effects of RP are most robust when retrieval is effortful, successful and spaced over time <sup>48,49</sup>. If retrieval of a learned item is practiced shortly after it is learned, but before it is forgotten, subsequent recall is enhanced, a phenomenon known as the "testing effect"<sup>47</sup>. RP has been used recently to improve performance of memory-impaired patients with multiple sclerosis<sup>50</sup> and M-STBI<sup>11,19</sup>.
- 6.2.4.1. <u>Procedure</u>. Six biweekly sessions of RP will be conducted. We will follow procedures outlined in Sumkowski et al<sup>19</sup>, who demonstrated efficacy of RP in a small group of patients with M-STBI and chronic memory deficits. For each session, two sets of 12 VPA's and 12 FNP's will be used. Paired stimuli will be presented together for 6s on a computer screen, and the participant will be asked to read the VPA or say the name (FNP) aloud. Following this, 3 6s filler pairs (other VPA's or FNP's) will be presented. Then, a 5s cued

recall test (candle-\_\_\_\_\_), followed by a 1-s feedback screen (candle-table) will be presented, followed by another six 6s filler trials and another 5s cued recall test and 1s feedback. This continues until all 12 VPA's or FNP's are given. After VPA is complete, FNP is administered (counterbalanced). After a brief delay, the participant completes two separate delayed cued recall tests (VPA, FNP, counterbalanced). The procedure is repeated for the second set of VPA's and FNP's. Dependent measure: Percent correct scores on the delayed recall test for each of the two VPA and two FNP sets, recorded each session.

6.2.5 <u>Manualization and Fidelity Testing.</u> During Phase 1, session-by-session procedures, including instructions to therapists and patients, stimuli and stimulus presentation schedules, methods of data collection, and permissible procedural variations will be formalized into a treatment manual for each of the three interventions. Six Master's level therapists will be trained in all three interventions, and will practice administering them to volunteer participants. At the end of Phase 1, each therapist will administer each treatment to a Veteran participant with M-STBI. Each session will be video recorded for evaluation of treatment fidelity by the study team<sup>51,52</sup>, which will review session recordings and will rate the degree to which the therapist adhered to the following aspects of the protocol: communication of content to the participant (consent, rationale for treatment, instructions for engaging in training), accurate use of cues, selection of stimulus materials, recording of data, and adherence to designated treatment schedules. We will develop a rating sheet that provides feedback to therapists on their adherence to the manualized protocol<sup>53</sup>.

# 6.3. Phase 2: Patient Characterization and Classification

- 6.3.1. Participants. Veterans aged 25-65 who are post-deployment, having served in OIF, OEF, or OND, who meet criteria for moderate or severe TBI during deployment, are eligible to participate. Patients will meet the 2007 VA/DoD criteria<sup>54</sup>, supplemented by data from the VA TBI Identification Semi-Structured Interview<sup>55</sup>. All patients will have gone through Level I and II assessments with positive findings. Inclusion/Exclusion criteria: Primary inclusion criteria: M-STBI (blast and blunt),  $\geq$  6 months post-injury, no receptive aphasia (impairing ability to comprehend task instructions), able to participate in return visits. Primary exclusion criteria: No MRI contraindications, not claustrophobic, no current or past history of disabling Axis I psychiatric disorders (except for PTSD and depression), no active substance abuse, not pregnant.
- 6.3.2. <u>Procedure</u>. Phase 2 consists of three components. **First**, after informed consent is obtained, participants undergo **standardized neuropsychological screening** to characterize their neurocognitive deficits, enabling comparisons with other Veterans whose memory rehabilitation outcomes have been reported in the literature. **Second**, we will use an established neuropsychometric algorithm to **classify patients into process-specific groups** that locates their primary memory deficit at the encoding, consolidation, or retrieval stage. **Third**, we will conduct **high-resolution structural and resting state functional MRI (RS-fMRI)** to determine whether our group classification is associated with different neuroimaging signatures. In this pilot proposal, we will not evaluate pre-post structural or functional brain changes resulting from our interventions, though this will be a key feature of a subsequent MERIT proposal based on our preliminary outcomes here.
- 6.3.2.1. <u>Pre-Treatment Neuropsychological Screening</u>. Table 1 lists key neuropsychological measures. Participants will be offered \$50 for participation in neuropsychological screening.

| Domain | Measure |
|---|---|
| Effort | Test of Memory Malingering (TOMM) |
| Intelligence | North American Adult Reading Test (NAART) |
| | Wechsler Abbreviated Scale of Intelligence (WASI 2-subtest) |
| Memory | California Verbal Learning Test II (CVLT-II) |
| | Rey Complex Figure Test (Meyers version) – includes forced-choice |
| | effort measure |
| | Logical Memory, Visual Reproduction I, II (WMS-III LM, VR) |
| Attention | WAIS-III Subtests yielding Working Memory Index (WMI); WMS-R DS |
| Processing Speed | WAIS-III Subtests yielding Processing Speed Index |
| Frontal/Executive | Controlled Oral Word Association Test (COWAT) – FAS, Animal |
| | Fluency |
| | Delis-Kaplan Executive Function System -Tower Test (DKEFS-Tower) |
| | Trail Making Test |
| Motor Speed and | Finger Tapping Test (FTT) |
| Dexterity | Grooved Pegboard Test (GPT) |
| Emotional/Psychiatric | PTSD Checklist-Military (PCL-M) |
| | Beck Depression Inventory |

# 6.3.2.2. Classifying Participants into Process-Specific Groups

We aim to identify M-STBI patients whose injuries produce primary deficits in encoding/acquisition, consolidation/retention, or retrieval. While we expect that many patients may have some problems in more than one domain, many studies have concluded that memory problems after M-STBI are primarily rooted in one of these domains at the individual level<sup>5-7,56,57</sup>. Three studies<sup>4,7,58</sup> report distinct deficit patterns attributable to encoding, consolidation, and retrieval deficits using the CVLT<sup>59</sup>. Crosson et al<sup>7</sup> found that encoding deficits were marked by a high false positive (FP) rate and reduced hits on recognition, while consolidation deficits were marked by lower hit rates and lower FP (also see<sup>58</sup>). Curtiss et al<sup>56</sup>, using hierarchical clustering of CVLT and WMS-R variables, found three memory-impaired groups corresponding to acquisition/encoding, retention, and retrieval deficits. Millis and Ricker<sup>4</sup> used Delis'<sup>59</sup> six-factor solution of CVLT performance variance to identify patterns of verbal learning deficit after moderate-severe TBI. They found 4 identifiable clusters: a *Disorganized* type (n = 22; encoding deficit) who exhibited a haphazard learning style, elevated FP rate, reduced discriminability on recognition testing and increased susceptibility to proactive interference, an Active type (n = 15; retrieval deficit) who showed good semantic encoding, good acquisition rate, and disproportionate improvement on recognition (discriminability), a *Passive* type (n = 11; consolidation deficit) whose recall showed prominent serial position effects and rapid forgetting, and a Deficient type (n = 13; encoding deficit) who showed slow rate of learning, recency effects in free recall, and an excessively high FP rate on recognition. These results were subsequently replicated and extended<sup>3</sup>. We will use this classification scheme, summarized in Table 2. Deficient and Disorganized groups will be collapsed, as both suffer from encoding deficits. Characteristics of each class (encoding, consolidation, and retrieval) will be combined in multivariate fashion, creating a composite score. Participants will be assigned to the group corresponding to the most impaired composite score. We will also investigate other algorithms for classifying patients, with the goal of deriving the most accurate and stable method.

Table 2. Scheme for Classifying TBI patients into deficit categories.

| Deficit | Encoding Deficit | Consolidation<br>Deficit | Retrieval Deficit |
|---|---|---|---|
| Millis/Ricker/Deshpande<br>Grouping | Disorganized (I) Deficient (IV) | Passive (III) | Active (II) |
| CVLT Factor Score<br>Comparisons | Serial cluster <iii,<br>=II<br/>Primacy <iii, =ii<br="">Slope &lt; II, =III<br/>FR Intrus =II, III<br/>List B v. A <ii, =iii<="" td=""><td>Serial cluster &gt;I,IV,=III Primacy <i,ii,>II Slope =I,IV, <ii <iv,="II" a="I,III,IV&lt;/td" b="" fr="" intrus="" list="" v.=""><td>Serial cluster =I, &gt;III Primacy <iii, =i,iv="" slope="">I,III,IV FR Intrus <iii,=i,iv a="" b="" list="" v.="">I, =III,IV</iii,=i,iv></iii,></td></ii></i,ii,></td></ii,></iii,></iii,<br> | Serial cluster >I,IV,=III Primacy <i,ii,>II Slope =I,IV, <ii <iv,="II" a="I,III,IV&lt;/td" b="" fr="" intrus="" list="" v.=""><td>Serial cluster =I, &gt;III Primacy <iii, =i,iv="" slope="">I,III,IV FR Intrus <iii,=i,iv a="" b="" list="" v.="">I, =III,IV</iii,=i,iv></iii,></td></ii></i,ii,> | Serial cluster =I, >III Primacy <iii, =i,iv="" slope="">I,III,IV FR Intrus <iii,=i,iv a="" b="" list="" v.="">I, =III,IV</iii,=i,iv></iii,> |
| CVLT Performance Features | False pos >II,III<br>Recency >II,III<br>Recog Discrim<br><ii,iii< td=""><td>False pos <i,ii,iv 5="" <i="" <ii="" cluster="" discrim="" recency="" recog="" sdfr="" semantic="" trial="" v.="">II</i,ii,iv></td><td>Semantic cluster &gt;III,IV SDFR v. Trial 5 <iii,iv consist="" fr="">I,IV Total (1-5) &gt;I,IV List B &gt;I,IV</iii,iv></td></ii,iii<> | False pos <i,ii,iv 5="" <i="" <ii="" cluster="" discrim="" recency="" recog="" sdfr="" semantic="" trial="" v.="">II</i,ii,iv> | Semantic cluster >III,IV SDFR v. Trial 5 <iii,iv consist="" fr="">I,IV Total (1-5) &gt;I,IV List B &gt;I,IV</iii,iv> |

- 6.3.2.3. <u>Structural/Functional Neuroimaging</u>. A long-term goal of our research is to provide evidence of neuroplastic changes after memory interventions by documenting treatment-related change in structural integrity and functional brain connectivity. In this study, we will collect pretreatment MRI data to provide brain-based biomarkers of our 3-group classification. Participants will be offered \$50 for participation in each of two MRI acquisitions, once before treatment, and again 1 month post-treatemtn.
  - 6.3.2.3.1. Acquisition Protocol. The MRI acquisition protocol is outlined in Table 3.
- 6.3.2.3.2. Structural MRI. Our laboratory uses tractography and tract-based spatial statistics<sup>60,61</sup> along with reliable manual segmentation of memory-relevant grey matter structures to analyze structural damage after TBI. Fiber orientation is estimated using the Mixture of Wishart (MOW) distribution method<sup>62</sup>, capable of estimating fiber orientation in regions of crossing fibers. Tractography will be performed by seeding the whole brain with 64 uniformly-spaced seeds within each voxel. The tracking algorithm (based on FACT<sup>63</sup>) creates connectivity streamlines using single and multi-fiber directionality. ROI's of key brain networks are defined anatomically and connected by streamlines. The streamlines with structural region masks will create a graph from which network edge weight (NEW)<sup>64</sup> will be computed. NEW controls for ROI surface area, seeding density, and voxel volume, and is a measure of network connection strength independent of image resolution, fiber length, and ROI size. NEW provides a quantitative measure of network connections that will be used together with FA and measures of radial and axial diffusivity to quantify structural brain integrity.
- 6.3.2.3.3. Resting-State Functional MRI. RS-fMRI, which measures intrinsic BOLD fluctuations in the absence of an explicit task, evaluates the degree to which activity in structurally connected brain regions co-varies (i.e., increases or decreases together) during rest. We will focus on resting state network connections between inferior frontal and medial temporal areas (shown to be prominent neural substrate of successful encoding<sup>65,66</sup>) and other resting state networks, including default mode network (DMN), task-positive network (TPN), and

salience network (SN). The *DMN* consists of interconnected regions in the posterior cingulate cortex, medial and lateral parietal cortex, and medial prefrontal cortex, which show *deactivation* during active task conditions<sup>67</sup>. The *TPN*, centered on connections between medial and dorsal regions of the frontal and parietal lobes, becomes more activated when the brain is presented with an attentionally demanding task<sup>68</sup>; activity within this region during encoding is associated with accurate retrieval later on<sup>69</sup>. The *SN*, comprised of dorsal anterior cingulate and the bilateral insula, responds to salient events and provides interaction between cortical, limbic, and subcortical structures essential for learning<sup>70</sup>. M-STBI is associated with abnormalities in the DMN<sup>71-74</sup>, TPN<sup>73</sup>, and SN<sup>75</sup>. It has been suggested<sup>73</sup> that TBI disrupts the normal segregation of

| Table 3. MRI Protocol – UF AMRIS 3T Philips System; 32 Channel Head Coil<br>Total Scan Time = 43m 55s | | |
|---|---|---|
| Sequences | Purpose | Parameters |
| 3D T1 | Gray-white<br>matter<br>segmentation | 176 continuous slices, voxel=1mm³, TR/TE=7.0/3.2ms, flip angle=8°, FOV=240x240mm, matrix=240x240x176mm, time: 4m 34s |
| 3D FLAIR | Structural lesion identification, segmentation | 180 continuous slices, voxel=1mm³, TR/TE=8000/338ms, IR=2400ms, flip angle=90°, FOV=240x240mm, matrix= 240x240x180mm, time: 7m 12s |
| T2 | Brain extraction | 176 continuous slices, voxel=1mm <sup>3</sup> ; TR/TE=2500/363ms; FOV=240x240, flip angle=90°; matrix=240x240x165; time: 5m 27s |
| SWI | Micro-<br>hemorrhage<br>detection | Flow-compensated gradient echo; TR/TE1/ΔTE=59/8/6ms, FOV=240x192mm, flip angle=22°, matrix=240x192x170mm, voxel=1x1x2mm³, time = 5m 31s |
| HARDI | Fiber integrity, fiber modeling | 74 continuous slices, 64 directions (1000s/mm²), 6 directions (100/mm²), voxel=2mm³, TR/TE=4840/86ms, flip angle=90°, FOV=224x224mm, matrix=224x224x140mm, time: 13m 1s |
| RS-BOLD | Resting state functional connectivity | 36 slices, Single-shot EPI sequence, TR/TE=2500/30ms, flip angle=90°, FOV=252x252mm, matrix=72x72x36mm, slice thickness=3.5mm, voxel=3.5mm³, time: 8m 10s |

the DMN and TPN through white matter damage to large corticortical pathways<sup>76,77</sup> and through damage to pathways that link the SN with the DMN and TPN. Such abnormalities are related to memory dysfunction<sup>73</sup> and show experience-dependent improvements after memory training<sup>31,78</sup>.

Participants will be asked to keep still during the entire scan to minimize motion artifacts. During resting state recording, participants will be asked to close their eyes, relax their body and mind, but not to fall asleep or focus on any specific thought. Total Interdependence (TI; developed by Co-I Ding), will be used to quantify the functional connectivity between pairs of ROIs. Compared with Cross Correlation (CC), which exploits the covariance structures of zero-lag data but ignores temporal relations that extend beyond zero-lag, TI estimates the total amount of mutual information between the two extracted BOLD time series<sup>79</sup>. The statistical treatment of TI is similar to that applied CC estimates, but it has been shown that, by revealing additional temporal relationships not captured by CC, TI reproduces more precise task activated networks, and provides greater sensitivity in correctly deciding network membership<sup>79</sup>.

# 6.4. Phase 3: Initial Testing of Treatment Efficacy

6.4.1. <u>Overview</u>. In this phase, appropriately classified patients will be assigned to participate in two memory interventions, one matched to their primary deficit, the other

mismatched, in counterbalanced order. The overall framework is outlined in Table 4; shaded cells are "matched" conditions.

6.4.2. <u>Design</u>. The overall approach is a *multiple-subject Alternating Treatment Design*, effective for determining the relative efficacy of two treatments in a single individual<sup>80</sup>. One participant will be assigned to each treatment order in Table 4, such that 4 patients per classification group (12 total) will participate. Each participant will receive 1 matched and 1

**Table 4. Treatment Schedule** 

| | Treatment Strategy/Target | | | Treatment Orders (one |
|---|---|---|---|---|
| Memory Deficit | Memory<br>Strategy<br>Training (1) | Errorless<br>Learning (2) | Retrieval<br>Practice (3) | matched, one mismatched; counterbalanced) |
| Encoding | +/+ | +/- | +/- | 12, 13, 21, 31 |
| Consolidation | -/+ | +/+ | +/- | 21, 23, 12, 32 |
| Retrieval | -/+ | -/+ | +/+ | 31, 32, 13, 23 |

mismatched treatment, in counterbalanced order. Therapists will be blinded to patient classification.

Although this design is subject to multiple-treatment interference<sup>81</sup> (the notion that the effects of each of the interventions might be affected by the presence of another intervention), such



Figure 1. Hypothetical data of two patients, one with encoding deficit (blue), the other with retrieval deficit (red).

carryover effects are typically small and counterbalancing the order of treatments should further reduce treatment carryover<sup>80</sup>. The design permits comparison of treatment effects in conditions in which a treatment is given first vs. second. New methods for calculating treatment effect size and possible confounding factors are available<sup>82-85</sup>. *It is hypothesized that greater gains in memory will be seen in matched, as compared to unmatched, treatments.* This is illustrated by hypothetical data presented in Figure 1, where a patient with encoding deficits (blue) benefits more [greater elevation and slope] from memory strategy training than from retrieval practice, while the opposite pattern is seen

in the patient with retrieval deficits (red). Each treatment will be conducted twice weekly for 3 weeks (6 sessions). Thus, each participant's involvement in actual treatment will span 6 weeks (2 treatments). Participants will be offered \$20/session for participation as inconvenience cost and to help them defray travel expenses. We will conduct a 1-month follow-up at which time performance on proximal outcomes (performance on VPA and FNP tasks) and secondary outcomes (see below) will be evaluated.

#### 6.5. Secondary Outcome Measures

We will collect preliminary data on secondary outcome measures (Table 5) derived from the Interagency Traumatic Brain Injury Outcomes Workgroup recommendations<sup>86</sup>. Measures will be collected before treatment, immediately after the conclusion of each treatment (during the last treatment session), and 1 month after treatment has concluded. The \$50 paid to the participant to undergo post-treatment MRI scanning will also cover the collection of 1-month post-treatment secondary outcome measures, since they will be collected on the same day.

Table 5. Secondary Outcome Measures

| Domain | Purpose | Measure |
|---|---|---|
| Global Outcome | Summarize overall TBI impact | MPAI-4 |
| Memory Impairment | Characterize memory deficits | RAVLT, BVMT-R, Everyday<br>memory simulations from<br>EON-MEM <sup>a</sup> |
| Social Role Participation | Evaluate involvement and participation in life situations | CHART-SF |
| Self-reported and general Quality of Life | Perceived satisfaction and well-being | SWLS, QUOLIBRI |
| Patient Reported Outcomes | Evaluate outcome from patient evaluation perspective | PROMIS <sup>b</sup> and Neuro-QOL <sup>c</sup><br>Item Banks |

<sup>&</sup>lt;sup>a</sup>Address/Phone Number, News Article, Face-Name Learning simulations; <sup>b</sup>Applied Cognition-Abilities, Applied Cognition-General Concerns; <sup>c</sup>Executive Function, General Concerns

### 7. Possible Discomforts and Risks:

- 7.1 Risks Associated with MRI: Magnetic resonance imaging (MRI) is a procedure that allows doctors to look inside the body by using a scanner that sends out a strong magnetic field and radio waves. This procedure is used routinely for medical care and is very safe for most people, but you will be monitored during the entire MRI scan in case any problems occur. The risks of MRI are:
- The MRI scanner contains a very strong magnet. Therefore, you may not be able to have the MRI if you have any type of metal implanted in your body, for example, any pacing device (such as a heart pacer), any metal in your eyes, or certain types of heart valves or brain aneurysm clips. Someone will ask you questions about this before you have the MRI.
- There is not much room inside the MRI scanner. You may be uncomfortable if you do not like to be in closed spaces ("claustrophobia"). During the procedure, you will be able to talk with the MRI staff through a speaker system, and, in the event of an emergency, you can tell them to stop the scan.
- The MRI scanner produces a loud hammering noise, which has produced hearing loss in a very small number of patients. You will be given earplugs to reduce this risk.
- If you are a woman of childbearing potential, there may be unknown risks to the fetus. Therefore, before you can have the MRI, you must have a pregnancy test.
- 7.2 <u>Risks Associated with Memory/Cognitive Testing</u>: When undergoing memory and cognitive ability testing, there is the risk of fatigue and frustration while taking the tests. Our trained examiners attempt to provide frequent breaks and utilize techniques to minimize frustration.
- 7.3 <u>Risks Associated with Participation in the Memory Treatment Program</u>: There are no known risks associated with participating in the memory treatment program.
- 7.4 <u>Other Risks</u>: Other possible risks to you may include: Normal risk associated with travel to and from UF and VA facilities.

# 8. Possible Benefits:

Patients may or may not benefit from participating in this research study. This research tests the effectiveness of memory rehabilitation therapies for helping Veterans with TBI-related memory problems. Since we are testing these treatments, we do not know how effective they are. Each participant will be given at least two such therapies, which may bring some benefit in memory by teaching strategies for remembering new information. The patient may also gain a better understanding of the effects of brain injury on memory function.

Other nonparticipating patients may benefit from our increased understanding of patterns of memory difficulty after mild traumatic brain injury that might respond better to particular memory rehabilitation therapies. Once we understand these patterns, we can better match patients to effective treatments designed to alleviate memory dysfunction.

**9. Conflict of Interest:** None, other than the typical benefit the PI and Co-I's get from presenting or publishing research results.

#### 10. Literature Cited

- 1 Bauer, R. M., Reckess, G. Z., Kumar, A. & Valenstein, E. Amnesic Disorders. In *Clinical Neuropsychology* (eds K.M. Heilman & E. Valenstein) 504-579 (Oxford University Press. 2012).
- 2 Rosenbaum, S. B. & Lipton, M. L. Embracing chaos: the scope and importance of clinical and pathological heterogeneity in mTBI. *Brain Imaging Behav* **6**, 255-282, doi:10.1007/s11682-012-9162-7 (2012).
- Deshpande, S. A., Millis, S. R., Reeder, K. P., Fuerst, D. & Ricker, J. H. Verbal learning subtypes in traumatic brain injury: a replication. *J Clin Exp Neuropsychol* 18, 836-842, doi:10.1080/01688639608408306 (1996).
- 4 Millis, S. R. & Ricker, J. H. Verbal learning patterns in moderate and severe traumatic brain injury. *J Clin Exp Neuropsychol* **16**, 498-507, doi:10.1080/01688639408402661 (1994).
- 5 DeLuca, J., Schultheis, M. T., Madigan, N. K., Christodoulou, C. & Averill, A. Acquisition versus retrieval deficits in traumatic brain injury: implications for memory rehabilitation. *Arch Phys Med Rehab* **81**, 1327-1333, doi:10.1053/apmr.2000.9390 (2000).
- Vanderploeg, R. D., Donnell, A. J., Belanger, H. G. & Curtiss, G. Consolidation deficits in traumatic brain injury: The core and residual verbal memory defect. *J Clin Exp Neuropsychol*, doi:10.1080/13803395.2013.864600 (2013).
- 7 Crosson, B., Novack, T. A., Trenerry, M. R. & Craig, P. L. California Verbal Learning Test (CVLT) performance in severely head-injured and neurologically normal adult males. *J Clin Exp Neuropsychol* **10**, 754-768, doi:10.1080/01688638808402812 (1988).
- 8 Vakil, E. The effect of moderate to severe traumatic brain injury (TBI) on different aspects of memory: a selective review. *J Clin Exp Neuropsychol* **27**, 977-1021, doi:10.1080/13803390490919245 (2005).
- 9 Stringer, A. Y. Ecologically-oriented neurorehabilitation of memory: robustness of outcome across diagnosis and severity. *Brain Injury : [BI]* **25**, 169-178, doi:10.3109/02699052.2010.541894 [doi] (2011).

- 10 Middleton, E. L. & Schwartz, M. F. Errorless learning in cognitive rehabilitation: a critical review. *Neuropsychol Rehabil* **22**, 138-168, doi:10.1080/09602011.2011.639619 [doi] (2012).
- 11 Sumowski, J. F., Coyne, J., Cohen, A. & Deluca, J. Retrieval practice improves memory in survivors of severe traumatic brain injury. *Arch Phys Med Rehab* **95**, 397-400, doi:10.1016/j.apmr.2013.10.021 (2014).
- 12 Belanger, H. G., Curtiss, G., Demery, J. A., Lebowitz, B. K. & Vanderploeg, R. D. Factors moderating neuropsychological outcomes following mild traumatic brain injury: a meta-analysis. *J Int Neuropsychol Soc: JINS* **11**, 215-227, doi:10.1017/s1355617705050277 (2005).
- 13 Wright, M. J. & Schmitter-Edgecombe, M. The impact of verbal memory encoding and consolidation deficits during recovery from moderate-to-severe traumatic brain injury. *J Head Trauma Rehab* **26**, 182-191, doi:10.1097/HTR.0b013e318218dcf9 (2011).
- 14 Wright, M. J., Schmitter-Edgecome, M. & Woo, E. Verbal memory impairment in severe closed head injury: the role of encoding and consolidation. *J Clin Exp Neuropsychol* **32**, 728-736 (2010).
- 15 Cicerone, K. D. *et al.* Evidence-based cognitive rehabilitation: updated review of the literature from 2003 through 2008. *Arch Phys Med Rehab* **92**, 519-530, doi:10.1016/j.apmr.2010.11.015 (2011).
- 16 Campbell, L., Wilson, F. C., McCann, J., Kernahan, G. & Rogers, R. G. Single case experimental design study of Carer facilitated Errorless Learning in a patient with severe memory impairment following TBI. *NeuroRehabilitation* **22**, 325-333 (2007).
- 17 Landis, J. *et al.* Evaluation of the errorless learning technique in children with traumatic brain injury. *Arch Phys Med Rehab* **87**, 799-805, doi:10.1016/j.apmr.2006.02.017 (2006).
- 18 Sumowski, J. F., Coyne, J., Cohen, A. & Deluca, J. Retrieval practice improves memory in survivors of severe traumatic brain injury. *Arch Phys Med Rehab*, doi:10.1016/j.apmr.2013.10.021 (2013).
- 19 Sumowski, J. F. *et al.* Retrieval practice: a simple strategy for improving memory after traumatic brain injury. *J Int Neuropsychol Soc : JINS* **16**, 1147-1150, doi:10.1017/s1355617710001128 (2010).
- 20 Haslam, C., Hodder, K. I. & Yates, P. J. Errorless learning and spaced retrieval: how do these methods fare in healthy and clinical populations? *J Clin Exp Neuropsychol* **33**, 432-447, doi:10.1080/13803395.2010.533155 (2011).
- 21 Small, J. A. A new frontier in spaced retrieval memory training for persons with Alzheimer's disease. *Neuropsychol Rehab* **22**, 329-361, doi:10.1080/09602011.2011.640468 (2012).
- 22 Glisky, E. L. & Schacter, D. L. Extending the limits of complex learning in organic amnesia: computer training in a vocational domain. *Neuropsychologia* **27**, 107-120 (1989).
- 23 Glisky, E. L., Schacter, D. L. & Tulving, E. Learning and retention of computer-related vocabulary in memory-impaired patients: method of vanishing cues. *J Clin Exp Neuropsychol* **8**, 292-312, doi:10.1080/01688638608401320 (1986).
- 24 Geary, E. K., Kraus, M. F., Rubin, L. H., Pliskin, N. H. & Little, D. M. Verbal learning strategy following mild traumatic brain injury. *J Int Neuropsychol Soc : JINS* **17**, 709-719, doi:10.1017/s1355617711000646 (2011).
- 25 Vakil, E., Arbell, N., Gozlan, M., Hoofien, D. & Blachstein, H. Relative importance of informational units and their role in long-term recall by closed-head-injured patients and control groups. *J Consult Clin Psychol* **60**, 802-803 (1992).

Protocol IRB version 03.09.04 PI version 3/4/2019 11:41 AM

- 26 Balota, D. A., Duchek, J. M., Sergent-Marshall, S. D. & Roediger, H. L. Does expanded retrieval produce benefits over equal-interval spacing? Explorations of spacing effects in healthy aging and early stage Alzheimer's disease. *Psychol Aging* **21**, 19-31 (2006).
- 27 Tulving, E. & Thompson, D. M. Encoding specificity and retrieval processes in episodic memory. *Psychol Rev* **80**, 352-373 (1973).
- 28 Nelson, D. L., McEvoy, C. L. & Schreiber, T. A. University of South Florida word association, rhyme, and word fragment norms. (1998). Downloaded 2/5/14 from <a href="http://www.usf.edu/FreeAssociation">http://www.usf.edu/FreeAssociation</a>.
- 29 Stringer, A. Y. *Ecologically Oriented Neurorehabilitation of Memory (EON-MEM)*. (Western Psychological Services, 2007).
- 30 Gross, A. L. & Rebok, G. W. Memory training and strategy use in older adults: results from the ACTIVE study. *Psychol Aging* **26**, 503-517, doi:10.1037/a0022687 (2011).
- 31 Hampstead, B. M., Stringer, A. Y., Stilla, R. F., Giddens, M. & Sathian, K. Mnemonic strategy training partially restores hippocampal activity in patients with mild cognitive impairment. *Hippocampus* **22**, 1652-1658, doi:10.1002/hipo.22006 (2012).
- 32 Shimamura, A. P. Episodic retrieval and the cortical binding of relational activity. *Cogn Affect Behav Neurosci* **11**, 277-291 (2011).
- 33 Addis, D. R. & McAndrews, M. P. Prefrontal and hippocampal contributions to the generation and binding of semantic associations during successful encoding. *Neuroimage* **33**, 1194-1206, doi:10.1016/j.neuroimage.2006.07.039 (2006).
- 34 Davachi, L. Item, context and relational episodic encoding in humans. *Cur Opin Neurobiol* **16**, 693-700, doi:10.1016/j.conb.2006.10.012 (2006).
- 35 Monti, J. M. *et al.* History of mild traumatic brain injury is associated with deficits in relational memory, reduced hippocampal volume, and less neural activity later in life. *Front Aging Neurosci* **5**, 41, doi:10.3389/fnagi.2013.00041 (2013).
- 36 Buckner, R. L. Functional-anatomic correlates of control processes in memory. *J Neurosci* **15**, 3999-4004 (2003).
- 37 Halford, G. S., Wilson, W. H. & Phillips, S. Relational knowledge: the foundation of higher cognition. *Trends Cogn Sci* **14**, 497-505, doi:10.1016/j.tics.2010.08.005 (2010).
- 38 Addis, D. R., Giovanello, K. S., Vu, M. A. & Schacter, D. L. Age-related changes in prefrontal and hippocampal contributions to relational encoding. *Neuroimage* **84**, 19-26, doi:10.1016/j.neuroimage.2013.08.033 (2014).
- 39 Hampstead, B. M., Sathian, K., Moore, A. B., Nalisnick, C. & Stringer, A. Y. Explicit memory training leads to improved memory for face-name pairs in patients with mild cognitive impairment: results of a pilot investigation. *J Int Neuropsychol Soc : JINS* **14**, 883-889, doi:10.1017/s1355617708081009 (2008).
- 40 Kessels, R. P. & de Haan, E. H. Implicit learning in memory rehabilitation: a meta-analysis on errorless learning and vanishing cues methods. *J Clin Exp Neuropsychol* **25**, 805-814, doi:10.1076/jcen.25.6.805.16474 (2003).
- 41 Anderson, N. D. & Craik, F. I. The mnemonic mechanisms of errorless learning. *Neuropsychologia* **44**, 2806-2813, doi:10.1016/j.neuropsychologia.2006.05.026 (2006).
- 42 Page, M., Wilson, B. A., Shiel, A., Carter, G. & Norris, D. What is the locus of the errorless-learning advantage? *Neuropsychologia* **44**, 90-100, doi:10.1016/j.neuropsychologia.2005.04.004 (2006).
- 43 Anderson, N. D., Guild, E. B., Cyr, A.-A., Roberts, J. & Clare, L. Contributions of frontal and medical temporal lobe functioning to the errorless learning advantage. *Neuropsychol Rehabil* **22**, 169-186 (2012).
- 44 Hunkin, N. M., Squires, E. J., Parkin, A. J. & Tidy, J. A. Are the benefits of errorless learning dependent on implicit memory? *Neuropsychologia* **36**, 25-36 (1998).

- 45 Clare, L. & Jones, R. S. Errorless learning in the rehabilitation of memory impairment: a critical review. *Neuropsychol Rev* **18**, 1-23, doi:10.1007/s11065-008-9051-4 (2008).
- 46 Pitel, A. L. *et al.* Two case studies in the application of errorless learning techniques in memory impaired patients with additional executive deficits. *Brain Injury : [BI]* **20**, 1099-1110, doi:10.1080/02699050600909961 (2006).
- 47 Roediger, H. L. & Karpicke, J. D. The power of testing memory: Basic research and implications for educational practice. *Perspectives on Psychological Science* **1**, 181-210 (2006).
- 48 Bjork, R. A. in *Metacognition: Knowing about knowing* (eds J. Metcalfe & A. Shimamura) 185-205 (MIT Press, 1994).
- 49 Cepeda, J. J., Pashler, H., Vul, E., Wixted, J. T. & Rohrer, D. Distributed practice in verbal recall tasks: A review and quantitative synthesis. *Psychol Bull* **132**, 354-380 (2006).
- 50 Sumowski, J. F., Chiaravalloti, N. & Deluca, J. Retrieval practice improves memory in multiple sclerosis: clinical application of the testing effect. *Neuropsychology* **24**, 267-272, doi:10.1037/a0017533 (2010).
- 51 Hart, T. & Bagiella, E. Design and implementation of clinical trials in rehabilitation research. *Arch Phys Med Rehab* **93**, S117-126, doi:10.1016/j.apmr.2011.11.039 (2012).
- 52 Persch, A. C. & Page, S. J. Protocol development, treatment fidelity, adherence to treatment, and quality control. *Amer J Occup Ther* **67**, 146-153, doi:10.5014/ajot.2013.006213 (2013).
- 53 Di Rezze, B., Law, M., Eva, K., Pollock, N. & Gorter, J. W. Development of a generic fidelity measure for rehabilitation intervention research for children with physical disabilities. *Devel Med Child Neurol* **55**, 737-744, doi:10.1111/dmcn.12114 (2013).
- 54 Assistant Secretary of Defense. *Traumatic Brain Injury: Definition and Reporting.* Washington DC: Department of Defense (2007).
- 55 Vanderploeg, R. D., Groer, S. & Belanger, H. G. Initial developmental process of a VA semistructured clinical interview for TBI identification. *JRRD* **49**, 545-555 (2012).
- 56 Curtiss, G., Vanderploeg, R. D., Spencer, J. & Salazar, A. M. Patterns of verbal learning and memory in traumatic brain injury. *J Int Neuropsychol Soc : JINS* **7**, 574-585 (2001).
- 57 Vanderploeg, R. D., Crowell, T. A. & Curtiss, G. Verbal learning and memory deficits in traumatic brain injury: encoding, consolidation, and retrieval. *J Clin Exp Neuropsychol* **23**, 185-195, doi:10.1076/jcen.23.2.185.1210 (2001).
- 58 Haut, M. W. & Shutty, M. S. Patterns of verbal learning after closed-head injury. *Neuropsychology* **6**, 51-58 (1992).
- 59 Delis, D. C., Kramer, J. H., Kaplan, E. & Ober, B. *California Verbal Learning Test Second Edition*. (Psychological Corporation, 2000).
- 60 Liu, Y. *et al.* Diffusion tensor imaging and Tract-Based Spatial Statistics in Alzheimer's disease and mild cognitive impairment. *Neurobiol Aging* **32**, 1558-1571, doi:S0197-4580(09)00336-4 [pii] 10.1016/j.neurobiolaging.2009.10.006 [doi] (2011).
- 61 Wada, T., Asano, Y. & Shinoda, J. Decreased fractional anisotropy evaluated using tract-based spatial statistics and correlated with cognitive dysfunction in patients with mild traumatic brain injury in the chronic stage. *AJNR Am J Neuroradiol* **33**, 2117-2122, doi:10.3174/ajnr.A3141 (2012).
- 62 Jian, B. & Vermuri, B. Milti-fiber reconstruction from diffusion MRI using mixture of wisharts and sparse deconvolution. *Inf Process Med Imaging* **20**, 384-395 (2007).
- 63 Mori, S., Crain, B., Chacko, V. & vanZihl, P. Three dimensional tracking of axonal projections in the brain by magnetic resonance imaging. *Ann Neurol* **45** (1999).

IRB version 03.09.04 PI version 3/4/2019 11:41 AM

- 64 Colon-Perez, L. et al. in International Society of Magnetic Resonance in Medicine. 2029 (Proc Intl Soc Mag Reson Med).
- 65 Diamond, E. L. *et al.* Relationship of fMRI activation to clinical trial memory measures in Alzheimer disease. *Neurology* **69**, 1331-1341 (2007).
- 66 Sperling, R. Functional MRI studies of associative encoding in normal aging, mild cognitive impairment, and Alzheimer's disease. *Ann N Y Acad Sci* **1097**, 146-155 (2007).
- 67 Raichle, M. E. & Snyder, A. Z. A default mode of brain function: a brief history of an evolving idea. *Neuroimage* **37**, 1083-1090; discussion 1097-1089, doi:10.1016/j.neuroimage.2007.02.041 (2007).
- 68 Fox, M. D. *et al.* The human brain is intrinsically organized into dynamic, anticorrelated functional networks. *Proc Natl Acad Sci U S A* **102**, 9673-9678 (2005).
- 69 Kim, H., Daselaar, S. M. & Cabeza, R. Overlapping brain activity between episodic memory encoding and retrieval: roles of the task-positive and task-negative networks. *Neuroimage* **49**, 1045-1054, doi:10.1016/j.neuroimage.2009.07.058 (2010).
- 70 Ham, T. E., Leff, A., De Boissezon, X., Joffe, A. & Sharp, D. J. Cognitive control and the salience network: An investigation of error processing and effective connectivity. *J Neurosci* **33**, 7091-7098 (2013).
- 71 Graner, J., Oakes, T. R., French, L. M. & Riedy, G. Functional MRI in the investigation of blast-related traumatic brain injury. *Front Neurol* **4**, 16, doi:10.3389/fneur.2013.00016 (2013).
- 72 Mayer, A. R., Mannell, M. V., Ling, J., Gasparovic, C. & Yeo, R. A. Functional connectivity in mild traumatic brain injury. *Hum Brain Mapp* **32**, 1825-1835, doi:10.1002/hbm.21151 (2011).
- 73 Sours, C. *et al.* Default mode network interference in mild traumatic brain injury a pilot resting state study. *Brain Res* **1537**, 201-215, doi:10.1016/j.brainres.2013.08.034 (2013).
- 74 Zhou, Y. *et al.* Default-mode network disruption in mild traumatic brain injury. *Radiology* **265**, 882-892, doi:10.1148/radiol.12120748 (2012).
- 75 Bonnelle, V. *et al.* Salience network integrity predicts default mode network function after traumatic brain injury. *Proc Natl Acad Sci U S A*, doi:10.1073/pnas.1113455109 (2012).
- 76 Niogi, S. N. & Mukherjee, P. Diffusion tensor imaging of mild traumatic brain injury. *J Head Trauma Rehab* **25**, 241-255, doi:10.1097/HTR.0b013e3181e52c2a (2010).
- 77 Mac Donald, C. L. *et al.* Detection of blast-related traumatic brain injury in U.S. military personnel. *N Engl J Med* **364**, 2091-2100, doi:10.1056/NEJMoa1008069 (2011).
- 78 Hampstead, B. M. *et al.* Activation and effective connectivity changes following explicit-memory training for face-name pairs in patients with mild cognitive impairment: a pilot study. *Neurorehab Neural Repair* **25**, 210-222, doi:1545968310382424 [pii] 10.1177/1545968310382424 [doi] (2011).
- 79 Wen, X., Mo, J. & Ding, M. Exploring resting state functional connectivity with total interdependence. *Neuroimage* **60**, 1587-1595 (2012).
- 80 Barlow, D. H. & Hayes, S. C. Alternating treatments design: One strategy for comparing the effects of two treatments in a single subject. *J Appl Beh Anal* **12**, 199-210 (1979).
- 81 Campbell, D. T. & Stanley, J. C. *Experimental and quasi-experimental designs for research.*, (Houghton Mifflin 1963).
- 82 Parker, R. I. & Hagan-Burke, S. Useful effect size interpretations for single case research. *Behav Ther* **38**, 95-105, doi:10.1016/j.beth.2006.05.002 (2007).

- 83 Parker, R. I. & Vannest, K. An improved effect size for single-case research: nonoverlap of all pairs. *Behav Ther* **40**, 357-367, doi:10.1016/j.beth.2008.10.006 (2009).
- 84 Parker, R. I., Vannest, K. J., Davis, J. L. & Sauber, S. B. Combining nonoverlap and trend for single-case research: Tau-U. *Behav Ther* **42**, 284-299, doi:10.1016/j.beth.2010.08.006 (2011).
- 85 Rusch, F. R. & Kazdin, A. E. Toward a methodology of withdrawal designs for the assessment of response maintenance. *J Appl Behav Anal* **14**, 131-140, doi:10.1901/jaba.1981.14-131 (1981).
- 86 Wilde, E. A. *et al.* Recommendations for the use of common outcome measures in traumatic brain injury research. *Arch Phys Med Rehab* **91**, 1650-1660 e1617, doi:10.1016/j.apmr.2010.06.033 (2010).